CLINICAL TRIAL: NCT07138430
Title: The Effect of Virtual Reality on Patient Outcome in Coronary Angiography
Brief Title: The Effect of Virtual Reality on Patient Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HARUN ÜNAL (Other)
Responsible Party: Sponsor-Investigator, HARUN ÜNAL, investigator, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1903
Record Dates: First submitted 2025-07-24; First posted 2025-08-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Coronary Angiography (CAG)
Keywords: Coronary Angiography; Virtual Reality; Nursing
MeSH Terms: interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In this study, patients in the intervention group were informed about the coronary angiography procedure and the virtual reality application.
  Interventions: Other: intervention group
- Control Group (Placebo Comparator): Patients in this group received no other interventions during the coronary angiography procedure other than standard care and treatment.
  Interventions: Other: standard care and treatment.

INTERVENTIONS:
Other: intervention group — In this study, patients in the intervention group were informed about the coronary angiography procedure and the virtual reality application. After completing the "Patient Identifier Form," the "Visual Analog Scale," and the "State Anxiety Inventory" 20 minutes before the procedure, the patients were placed in the supine position in the procedure room to prepare for the procedure. Two minutes before the coronary angiography, the patients were fitted with virtual reality headsets, and throughout the procedure, they listened to images of nature, forests, and riverside areas, along with accompanying relaxing music. Twenty minutes after the procedure, the patients' pain, anxiety, and satisfaction levels were re-evaluated using the scales. One week after discharge, the patients were evaluated in the cardiology outpatient clinic for pain, hematoma, and edema in the femoral region, and the "Visual Analog Scale" was administered again.
  Arms: intervention group
Other: standard care and treatment. — The pre-procedure preparations for patients in the control group were similar to those in the intervention group. Patients in this group received no other interventions during the coronary angiography procedure other than standard care and treatment. Control group patients completed the VAS and anxiety scale 20 minutes after the procedure. Post-discharge procedures for the control group were identical to those for the intervention group.
  Arms: Control Group

SUMMARY:
This study explores the impact of virtual reality (VR) interventions on patient outcomes during coronary angiography procedures. It evaluates the effectiveness of VR in reducing patient anxiety, enhancing comfort, and improving overall satisfaction. The findings suggest that the use of VR as a non-pharmacological support tool can positively influence patients' emotional states, reduce perceived stress levels, and potentially improve cooperation during the procedure. These results highlight the potential of immersive technologies to support patient-centered care in interventional cardiology settings.

DETAILED DESCRIPTION:
Coronary angiography is an essential diagnostic and interventional procedure widely used to assess coronary artery disease. Despite its clinical importance, many patients experience significant levels of anxiety, stress, and discomfort before and during the procedure, which can negatively impact their physiological responses and overall satisfaction. In recent years, non-pharmacological interventions, particularly immersive technologies such as virtual reality (VR), have been investigated for their potential to enhance the patient experience during medical procedures.

This study aimed to evaluate the effect of virtual reality on patient outcomes during coronary angiography. A controlled clinical trial design was employed to compare a group of patients exposed to a VR intervention-typically involving calming, immersive environments-against a control group receiving standard care. Key outcome measures included anxiety levels, pain perception, and overall patient satisfaction.

The study supports the integration of virtual reality as a complementary tool in cardiac catheterization laboratories to improve patient-centered outcomes. As technology becomes increasingly accessible, VR-based interventions may offer innovative solutions to reduce procedural stress and improve the quality of care in invasive cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70,
* Who volunteer to participate in the study,
* Who are open to communication, who can read and write,
* Patients without visual or auditory impairments,
* Patients who have undergone femoral artery bypass grafting,
* Patients who have not received opioids or tranquilizers,
* Patients undergoing coronary angiography for the first time will be included in the study.

Exclusion Criteria:

* Patients who have difficulty using virtual reality glasses and who experience headaches, nausea, and vomiting
* Patients under the age of 18
* Pregnant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | 10 minutes
  Description: This form, prepared by researchers based on literature review, consists of a total of 11 questions to question the socio-demographic characteristics and disease-related characteristics of patients.
Visual Analog Scale | 10 minutes
  The VAS, whose validity and reliability study was conducted by Price et al. (1983), is a tool that subjectively assesses and measures people's pain experiences. The VAS is frequently used in assessing pain levels in adults and is considered the fastest and simplest to understand among single-dimensional scales. To determine pain intensity, the patient is asked to mark the score corresponding to the quantitative pain experienced on a 10-cm ruler, with the "0" point at one end representing "no pain" and the "10" point at the other end representing "the most severe pain." The scale can be applied horizontally or vertically. The point marked by the patient is used as numerical data to determine the level of pain perception. On this scale, a "0" point indicates no pain, while a "10" point describes the most severe pain.
State Anxiety Scale | 10 minutes
  Description: The study used the "State and Trait Anxiety Scale," developed by Spielberger et al. (1970) and translated and adapted into Turkish by Öner and Le Compte (1998). The scale consists of a total of 40 items and two separate scales. The first section includes the "State Anxiety Scale," which measures how a person feels at a specific moment, and the second section includes the "Trait Anxiety Scale," which includes statements about how a person feels in general. This study was designed for use during coronary angiography, and the "State Anxiety Scale" was used based on a literature review and expert opinions.
SATISFACTION EVALUATION SCALE | 5 minutes
  SATISFACTION EVALUATION SCALE Please indicate your level of satisfaction with the use of virtual reality headsets on a scale between 0 (zero) and 10 (ten).

CONTACTS AND LOCATIONS:
Locations (1):
- Van YYÜ Univercity, Van, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided